CLINICAL TRIAL: NCT03285542
Title: Prospective Randomized Trial of Dermabond Prineo Wound Closure System on Operating Room Time and Wound Closure Time in Total Knee Arthroplasty
Brief Title: Prospective Randomized Trial of Dermabond Prineo in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Viktor Krebs, M.D., Vice Chairman - Adult Reconstruction, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-842
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Wound Heal
Keywords: adhesive; total knee arthroplasty; wound; closure; time; barbed suture; knoteless suture
MeSH Terms: conditions — Wounds and Injuries | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DERMABOND GROUP (Active Comparator): For the active arm of the study, the arthrotomy (deep layer) is repaired using number 1 Vicryl, the subcutaneous layer will be then closed with simple interrupted knots using number 2-0 braided absorbable sutures (Vicryl), followed by closure of the subcutaneous layer using a STRATAFIX Spiral Knotless Tissue Control Device in addition to DERMABOND PRINEO (Ethicon, Johnson and Johnson, Somerville, New Jersey) system for dermal closure.
  Interventions: Device: DERMABOND
- CONTROL GROUP (Placebo Comparator): For the control arm of the study, the arthrotomy (deep layer) is repaired using number 1 Vicryl, the subcutaneous layer will be then closed with simple interrupted knots using number 2-0 braided absorbable sutures (Vicryl), followed by skin closure with staples
  Interventions: Device: Staples

INTERVENTIONS:
Device: DERMABOND — DERMABOND PRINEO (Ethicon, Johnson and Johnson, Somerville, New Jersey)
  Arms: DERMABOND GROUP
Device: Staples — staples for skin closure
  Arms: CONTROL GROUP

SUMMARY:
In this prospective pilot study examining the superficial closure during total knee arthroplasty, active subjects will receive the STRATAFIX Spiral Knotless Tissue Control Device for subcuticular closure in addition to DERMABOND PRINEO (Ethicon, Johnson and Johnson, Somerville, New Jersey) system for dermal closure. The control subjects will receive staples (standard-of-care).

DETAILED DESCRIPTION:
The DERMABOND PRINEO (Ethicon, Johnson and Johnson, Somerville, New Jersey) system is a unique two-part skin closure system that consists of: a 2-octyl cyanoacrylate topical skin adhesive for proven strength and microbial protection in vitro, and a flexible, self-adhesive polyester mesh for excellent approximation and healing. It is aimed to add strength and protection when closing medium to long incisions. In addition, it is designed to replace the use of subcuticular sutures or staples, with greater holding strength, with the potential to reduce skin closure time.

Various studies have evaluated the outcomes of different closure devices, however, there are no reports assessing the length of closure times using DERMABOND PRINEO (Ethicon, Johnson and Johnson, Somerville, New Jersey) Knotless Tissue Control Devices during superficial closure in orthopaedic surgery. Huemer et al. (1) performed an observational study of 180 patients who had 224 excisional body-contouring surgeries utilizing Dermabond Prineo for superficial closure. Authors concluded that this closure type enables the surgeon to perform a quick and smooth skin closure. However, 4 patients (1.8%) developed local allergic reactions, which necessitated early removal and topical corticosteroid treatment. Parvizi et al.(2) performed an open, prospective, randomized clinical study of superficial wound closure on 60 patients undergoing abdominoplasty with either Dermabond Prineo or conventional superficial closure. They found significantly lower price ($134.79 cheaper) and significantly better Hollander Cosmesis Scale scores in Dermabond Prineo cohort. In addition, there was a significantly better cosmetic outcome at 6 and 12 months after surgery. The use of Dermabond Prineo may be able to decrease operative time and costs in other surgical fields, such as orthopedics. Careful patient allergy history is necessary to avoid adhesive allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, between the ages of 18 to 80 years at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Able to fluently speak and understand the local language
5. If female, is nonpregnant (negative pregnancy test results at the baseline/randomization visit) and nonlactating.
6. End-stage osteoarthritis patients planning to undergo primary total knee arthroplasty
7. BMI less than 40 kg/m2

Exclusion Criteria:

1. BMI greater than or equal to 40 kg/m2
2. History of known bleeding disorder
3. History of medical co-morbidity that may result in poor wound healing (ie. diabetes mellitus, peripheral vascular disease)
4. Patients <18 or >80 years of age
5. Patients who are prisoners
6. Mentally unable to sign informed consent
7. Has an uncontrolled illness that, in the opinion of the investigator, is likely to cause the patient to be withdrawn from the trial or would otherwise interfere with interpreting the results of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Krebs, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DERMABOND GROUP | CONTROL GROUP
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DERMABOND GROUP | CONTROL GROUP | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 62 (7) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 8 | 15 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Modified Hollander Cosmesis Scale
Description: Scar evaluation scale is used to assess the long-term aesthetic or cosmetic appearance of scars.
  Scars were assigned 0 or 1 point each for the presence (1) or absence (0) of the following: (1) a width greater than 2 mm at any point of the scar; (2) a raised or depressed scar in relation to the surrounding normal skin; (3) red, blue, brown, or black discoloration of the scar relative to the surrounding normal skin; (4) any hatch marks on either side of the scar from previous sutures or staples; and (5) overall poor or ugly appearance. The total score was then derived by adding the scores on the individual items of the scar evaluation scale ranging from 0 (best) to 5 (worst).
Time Frame: 90 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | DERMABOND GROUP | CONTROL GROUP
Number analyzed (Participants) | 30 | 30
Participants
  Total score 0 | 30 | 0
  Total score 1 | 0 | 23
  Total score 2 | 0 | 5
  Total score 3 | 0 | 1
  Total score 4 | 0 | 1
  Total score 5 | 0 | 0

2. Secondary Outcome: Number of Patients With Wound Complications
Description: presence of superficial wound infection, deep wound infection, periprosthetic joint infection, wound hematoma, and wound dehiscence.
Time Frame: 90 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | DERMABOND GROUP | CONTROL GROUP
Number analyzed (Participants) | 30 | 30
Participants | 2 | 0

3. Secondary Outcome: Patient Satisfaction (Visual Analogue Scale)
Description: patient satisfaction with wound appearance, measured by marking on a line of 100 mm, with 0 mm being low and 100 mm being high.
Time Frame: 90 days postoperative
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | DERMABOND GROUP | CONTROL GROUP
Number analyzed (Participants) | 30 | 29
millimeters | 97.6 (3.2) | 82.6 (12.8)

ADVERSE EVENTS:
Time Frame: 90 days postoperative
Arm/Group | DERMABOND GROUP | CONTROL GROUP
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DERMABOND GROUP (N=30) | CONTROL GROUP (N=30)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Superficial surgical site infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03285542/Prot_SAP_000.pdf